CLINICAL TRIAL: NCT03502044
Title: New MRT Imaging Biomarkers and Treatment With Kinetic Oscillatory Stimulation (KOS) in Nasal Cavity for Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Tie-Qiang Li, Adjunct Professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KarolinskaUH2018
Record Dates: First submitted 2018-03-23; First posted 2018-04-18 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Myalgic Encephalomyelitis; Chronic Fatigue Syndrome
Keywords: Myalgic Encephalomyelitis; Chronic Fatigue Syndrome; Kinetic Oscillatory Stimulation in nasal cavity
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Intervention Model Description: Double blinded placebo controlled trial design during the first 8 treatments. Single blinded (patient is blinded) controlled trial design during the last 8 treatments.
Who Masked: Participant, Investigator
Masking Description: Both the participants and investigator are blinded with regarding the administration of KOS or placebo treatments during the first 8 treatments.
  During the following 8 treatments only the patients, not the investigator, are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1, active KOS treatment (Active Comparator): Patients in arm 1 receive active KOS treatment throughout study, which means 16 active KOS treatments. Patients receive KOS treatments twice a week during 8 consecutive weeks.
  Interventions: Device: Active Kinetic Oscillation Stimulation (KOS)
- Arm 2, 8 inactive KOS treatments then 8 active KOS treatments (Placebo Comparator): Patients in arm 2 receive inactive KOS treatment during the first 8 KOS treatments of the study. Thereafter patients in arm 2 receive 8 active KOS treatments. Patients receive KOS treatments twice a week during 8 consecutive weeks.
  Interventions: Device: Inactive Kinetic Oscillation Stimulation (KOS); Device: Active Kinetic Oscillation Stimulation (KOS)

INTERVENTIONS:
Device: Inactive Kinetic Oscillation Stimulation (KOS) — 10 minutes inactive KOS treatment in each nasal cavity.
  Arms: Arm 2, 8 inactive KOS treatments then 8 active KOS treatments
Device: Active Kinetic Oscillation Stimulation (KOS) — 10 minutes active KOS treatment in each nasal cavity.

SUMMARY:
Placebo controlled trial study of efficacy of Kinetic Oscillation Stimulation (KOS) in nasal cavity will be conducted in patients with myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS). The outcome of the treatment will be assessed with clinical evaluation of patients, cognitive tests, structural and functional MRI of the brain.

DETAILED DESCRIPTION:
Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS) is a neurologic disease that is characterized by extreme physical and mental fatigue. Although some signs of inflammation have been reported previously in ME/CFS patients, the data have been quite limited and controversial. A recent study based on multiplex array of a Luminex system has demonstrated an immune signature of serum cytokines that is correlated with the disease severity and fatigue duration. Results from resting-state functional MRI (fMRI) studies have also demonstrated that there is a significant correlation between the degree of chronic fatigue and reduction of functional network connectivity in the brain.

The autonomic nervous system (ANS) plays an important role in the regulation of systemic inflammation. The nasal cavity has a rich innervation of cranial nerves. We have recently developed a non-invasive ANS stimulation technique, called Kinetic Oscillation Stimulation (KOS) in the nasal cavity. KOS treatment is expected to have a positive impact on systemic inflammation via the restoration of ANS homeostasis.

With this double blinded, placebo controlled, clinical trial, the efficacy of KOS treatment on ME/CFS will be assessed by clinical evaluation, multiplex immunoassay of peripheral blood samples, performance of psychomotor vigilance task, structural and functional MRI of the brains at the baseline point before KOS treatment and after the completion of KOS treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS) established by Consultant in Neurology.

Exclusion Criteria:

* Any cardiovascular disease.
* Any other condition considered by the physician to render the patient unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-06-15 (Estimated)

PRIMARY OUTCOMES:
Change in Fatigue severity scale | Baseline before KOS intervention, immediately after every second KOS treatment, 3 months after last KOS treatment.
  A 9-item questionnaire with questions related to how fatigue interferes with certain activities and rates its severity according to a self-report scale. The items are scored on a 7 point scale with 1 = strongly disagree and 7= strongly agree. Maximum score possible is 63.

SECONDARY OUTCOMES:
Diagnostic MRI of the brain | At baseline before KOS intervention and within 4 weeks after the last KOS intervention (16 KOS interventions are given during 8 consecutive weeks)
  Functional MRI of the brain at 3T
Signature of systemic inflammation and severity | At baseline before KOS intervention and within 4 weeks after the last KOS intervention (16 KOS interventions are given during 8 consecutive weeks)
  Analysis of high dimensional immune signature from peripheral venous blood samples using mass cytometry.
SF-36 PHYSICAL FUNCTIONING SUBSCALE (PF-10) SF-36 Physical Functioning Subscale (PF-10) | At baseline before KOS intervention, immediately after 8 treatments, immediately after 16 treatments, 3 months after the last treatment.
  The PF-10 is a generic outcome measure designed to examine a person's perceived limitation with physical functioning and is a subscale within the Medical Outcomes Study 36-item Short Form Health Survey (SF-36). There are 10 items, each item is rated on a 3-point scale.
ME/CFS symptom rating scale | At baseline before KOS intervention, immediately after every second KOS treatment, 3 months after last KOS treatment.
  Series of questions regarding ME/CFS symptoms graded 0-5 to evaluate degree of disease burden, according to the diagnostic Canadian Criteria.
Hospital anxiety depression scale (HADS) | At baseline before KOS intervention, immediately after 8 treatments, immediately after 16 treatments, 3 months after the last treatment.
  The questionnaire comprises 7 questions for anxiety and 7 questions for depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.

CONTACTS AND LOCATIONS:
Overall Officials: Per Julin, MD, PhD, Study Director — Neurological Rehabilitation Clinic in Stora Sköndal
Locations (1):
- Neurological Rehabilitation Clinic in Stora Sköndal, Stockholm, Sweden